CLINICAL TRIAL: NCT01774994
Title: Arginine and Nitric Oxide (NO) Metabolism in Healthy Human Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Basic Science
Other Study IDs: MEC04-021.3
Record Dates: First submitted 2013-01-22; First posted 2013-01-24 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Healthy
Keywords: volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- stable isotopes (Experimental): stable isotope infusion for measurement of metabolism
  Interventions: Other: stable isotope infusion for measurement of metabolism

INTERVENTIONS:
Other: stable isotope infusion for measurement of metabolism

SUMMARY:
Investigation of arginine and NO metabolism in healthy subjects is important as a reference for alterations in arginine-NO metabolism in patients. Moreover, this study will indicate the changes during aging and gender-related differences. Although data on arginine metabolism exist in literature, data are limited to young healthy male subjects. Since patients with suspected changes in arginine metabolism, e.g. sepsis and cancer patients are often elderly and also women, knowledge of arginine metabolism in these groups is needed.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age 18-25 years (young); 50-70 years (middle aged/elderly)

Exclusion Criteria:

* Diabetes mellitus type I
* Livercirrhosis, pancreatitis, malignancies
* Hypertension (diastolic blood pressure >95 mmHg or systolic blood pressure >160 mmHg)
* History of gastrointestinal complaints
* Recent involuntary weight loss (more than 10 % in 6 months or more than 5 % in one month)
* Pregnancy (pregnancy test is done in female subjects)
* Use of medication that can affect arginine metabolism (nitrovasodilators and corticosteroids)
* Subjects with "high activity level"

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2004-11; Primary Completion 2005-01 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
whole body NO synthesis | 2 hours
  postabsorptive nitric oxide synthesis measured by using stable isotope methodology

SECONDARY OUTCOMES:
whole body protein metabolism | 2 hours
  postabsorptive whole body protein metabolism (protein synthesis, breakdown, net protein breakdown) measured by using stable isotope methodology
whole body arginine metabolism | 2 hours
  postabsorptive arginine metabolism measured by using stable isotope methodology
blood parameters | 2 hours
  postabsorptive blood levels (glucose, insulin, urea, amino acids, CRP)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaas E Deutz, MD PhD, Principal Investigator

REFERENCES:
- [Background] Luiking YC, Ten Have GA, Wolfe RR, Deutz NE. Arginine de novo and nitric oxide production in disease states. Am J Physiol Endocrinol Metab. 2012 Nov 15;303(10):E1177-89. doi: 10.1152/ajpendo.00284.2012. Epub 2012 Sep 25. PMID 23011059
- [Background] Luiking YC, Engelen MP, Deutz NE. Regulation of nitric oxide production in health and disease. Curr Opin Clin Nutr Metab Care. 2010 Jan;13(1):97-104. doi: 10.1097/MCO.0b013e328332f99d. PMID 19841582